CLINICAL TRIAL: NCT02436460
Title: A Phase Ib Treatment Trial Using AbGn-168H to Treat Steroid Refractory Acute Graft-vs.-Host Disease (aGVHD) in Patients Undergoing Allogeneic Hematopoietic Cell Transplantation
Brief Title: A Study of AbGn-168H in Patients With Steroid Refractory Acute Graft-vs-Host Disease After Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Re-initiate a new trial per the discussion with FDA
Sponsor: AbGenomics B.V Taiwan Branch (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 285; NCI-2015-00631 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-32842; 348; BMT 285 (Other: Stanford University Hospitals and Clinics)
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Acute Graft Versus Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AbGn-168H (Experimental): AbGn-168H will be administered once weekly for four weeks via intravenous infusion.
  Interventions: Biological: AbGn-168H

INTERVENTIONS:
Biological: AbGn-168H — Humanized monoclonal antibody
  Other Names: Neihulizumab

SUMMARY:
This study is to establish the safety, determine if there is an improvement in steroid refractory acute graft-vs-host disease (aGvHD) compared to historical cohorts, and determine the changes of aGvHD-associated T-cell clones in patients with steroid-refractory aGVHD following allogeneic hematopoietic cell transplantation administered AbGn-168H once weekly for 4 weeks.

DETAILED DESCRIPTION:
AbGn-168H is a humanized monoclonal antibody. This is a dose escalation study using a modified toxicity probability interval method. AbGn-168H will be administered intravenously (IV) once weekly for four weeks, in patients with steroid refractory aGVHD following hematopoietic cell transplant (HCT). After completion of study treatment, patients are followed up for 90 days.The primary objective of this study is to establish the safety, and the secondary objectives of this study are to determine if there is an improvement in disease response at 3 months after diagnosis of steroid refractory aGVHD compared to historical cohorts and to determine the changes in frequency and/or phenotype of aGVHD-associated T cell clones in response to AbGn-168H therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of skin, gut and/or liver steroid-refractory GVHD by clinical assessment of treating physician following allogeneic HCT. Patients who fail to respond to steroids by 7 days are considered steroid-refractory
2. Previously-treated with any conditioning regimen and any GVHD immune suppression prophylaxis and formulation of steroids, except as noted in Exclusion Criteria #2.
3. AbGn-168H (neihulizumab) therapy can begin not more than 14 days after diagnosis of aGvHD
4. Karnofsky Performance Status (KPS) > 50%
5. No evidence of HCT graft failure or multi-organ failure
6. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Uncontrolled infections not responsive to antimicrobial therapy requiring intensive critical care
2. Progressive malignant disease, including post-transplant lymphoproliferative disease unresponsive to therapy
3. Treatment with investigational GVHD prophylactic agents (eg, CCR5 inhibitors; lenalidomide; and/or bortezomib) within the 7 days prior to the 1st dose of neihulizumab
4. Treatment with other investigational agents within the prior 7 days prior to the 1st dose of AbGn-168H (neihulizumab)
5. CMV PCR > 500 copies/mL or evidence of end-organ damage due to CMV
6. Pregnant or nursing
7. HIV positivity (NOTE: patients positive for hepatitis B or hepatitis C are not excluded, and may be evaluated on a case-by-case basis)
8. Renal clearance CCR < 40 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Adverse events | On or before study day 52
  Grade 3 to 5 adverse events considered at least possibly-related to neihulizumab
Cytokine release syndrome or acute infusion reactions | Within 24 hours after study drug infusion
  Grade 3 to 5 cytokine release syndrome or acute infusion reactions
Neutropenia | Duration of study
  Grade 4 neutropenia lasting more than 14 days considered at least possibly related to study drug
All-cause mortality | Within 7 days of infusion
  Grade 5 all-cause mortality

SECONDARY OUTCOMES:
Changes in frequency and/or phenotype of aGVHD-associated T-cell clones | At time of diagnosis up to 90 days
  Changes in T cell clonal dynamics will be accomplished by statistical methodology.
GVHD treatment response as measured by the Modified Keystone aGVHD clinical grade scale | At 90 days after the diagnosis of aGVHD
  Treatment response will be estimated by the Kaplan Meier product limit method, with standard confidence limits

CONTACTS AND LOCATIONS:
Overall Officials: Shih-Yao (David) Lin, MD, PhD, Study Director — AbGenomics B.V.; Everett Meyer, MD, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No